CLINICAL TRIAL: NCT01270763
Title: Gene x Behavior Interaction in the Look AHEAD Study
Status: Completed | Type: Observational
Sponsor: The Miriam Hospital (Other)
Collaborators: Tufts Medical Center (Other); Brown University (Other)
Responsible Party: Principal Investigator, Jeanne McCaffery, Senior Research Scientist/Associate Professor, The Miriam Hospital
Other Study IDs: GxB in Look AHEAD
Record Dates: First submitted 2010-11-12; First posted 2011-01-05 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Obesity; physical fitness; cholesterol levels; genetics; weight loss
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Weight Loss | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA obtained as part of the parent study
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- The Look AHEAD Study: The Look AHEAD Study includes intensive lifestyle intervention treatment, focusing on caloric intake and physical activity, and a treatment arm focused on diabetes support and education.
  Interventions: Behavioral: Intensive lifestyle intervention; Behavioral: Diabetes support and education

INTERVENTIONS:
Behavioral: Intensive lifestyle intervention — Lifestyle intervention focused on weight loss through diet and physical activity
Behavioral: Diabetes support and education — Behavioral intervention focused on diabetes support and education

SUMMARY:
The interplay of genetic and behavioral factors is critical to understanding obesity. Behavioral weight loss intervention has emerged as a key strategy in combating obesity. However, individuals differ in their degree of success in these programs and genetic factors are known to play a role. In this application, the investigators propose to identify specific genes that predict individual differences in weight loss and high density lipoprotein cholesterol in response to behavioral intervention to help identify individuals that struggle with weight loss and cholesterol despite behavioral efforts.

DETAILED DESCRIPTION:
The interplay of genetic and behavioral factors is critical to understanding obesity. Obesity is a major public health problem, with millions of Americans suffering from weight-related health complications, including Type 2 diabetes, coronary heart disease, hypertension, and osteoarthritis. Behavioral weight loss intervention has emerged as a key strategy in combating obesity and the associated health consequences. However, individuals differ in their degree of success in these programs even if they make the recommended behavioral changes and genetic factors are known to play a role. In this application, the investigators propose to identify specific genes that predict individual differences in weight loss in response to behavioral intervention to help identify individuals who struggle with weight loss despite behavioral efforts. Specifically, the investigators will determine whether obesity genes interact with lifestyle intervention in predicting weight loss at year 1 of the Look AHEAD trial, an NIH-funded, multi-center randomized controlled trial with the primary goal of determining whether weight loss achieved through an intensive lifestyle intervention can reduce cardiovascular morbidity and mortality among persons with type 2 diabetes. At year 1, participants assigned to Intensive Lifestyle Intervention (ILI), focusing on changes in diet and physical activity, lost an average of 8.6% of their weight (N = 2,496; 97.1% follow-up) relative to losses of 0.7% among individuals assigned to the Diabetes Support and Education (DSE) group (N= 2,463, 95.7% follow-up), who received diabetes support and education groups alone. Consent for genetic analyses was provided by 3,759 participants. Genotype data from the IBC chip, a genotyping platform including 50,000 single nucleotide polymorphisms (SNPs) from ~2,600 genes relevant to cardiovascular disease, lipid metabolism, diabetes and obesity, will allow us to test the central hypothesis that genes that predispose to obesity interact with lifestyle treatment to influence weight loss following intensive lifestyle intervention. The investigators will also determine whether genes related to high density lipoprotein (HDL) cholesterol predict the degree of improvement in HDL in response to the behavioral intervention. The investigators conduct these aims with the explicit goal of bringing together a team with expertise in behavioral research, genetic epidemiology and molecular biology to create transdisciplinary researchers who are able to bridge across the disciplines and identify key gene x behavior interactions in the context of the Look AHEAD trial.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the Look AHEAD Study, genetic consent

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 5,145 individuals who are overweight or obese, have type 2 diabetes and are enrolled in the Look AHEAD Study
Sampling Method: Non-Probability Sample
Enrollment: 4108 (Actual)
Dates: Start 2009-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Body weight | 4 years
High density lipoprotein cholesterol | 4 years

SECONDARY OUTCOMES:
Dietary intake | 4 years
Physical activity/fitness | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne McCaffery, Ph.D., Principal Investigator — The Miriam Hospital; Rena Wing, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Look AHEAD Research Group. Prospective Association of GLUL rs10911021 With Cardiovascular Morbidity and Mortality Among Individuals With Type 2 Diabetes: The Look AHEAD Study. Diabetes. 2016 Jan;65(1):297-302. doi: 10.2337/db15-0890. Epub 2015 Sep 22. PMID 26395743
- [Derived] Look AHEAD Research Group. Prospective association of a genetic risk score and lifestyle intervention with cardiovascular morbidity and mortality among individuals with type 2 diabetes: the Look AHEAD randomised controlled trial. Diabetologia. 2015 Aug;58(8):1803-13. doi: 10.1007/s00125-015-3610-z. Epub 2015 May 14. PMID 25972230
- [Derived] McCaffery JM, Papandonatos GD, Huggins GS, Peter I, Erar B, Kahn SE, Knowler WC, Lipkin EW, Kitabchi AE, Wagenknecht LE, Wing RR; Genetic Subgroup of Look AHEAD; Look AHEAD Research Group. Human cardiovascular disease IBC chip-wide association with weight loss and weight regain in the look AHEAD trial. Hum Hered. 2013;75(2-4):160-74. doi: 10.1159/000353181. Epub 2013 Sep 27. PMID 24081232
- [Derived] McCaffery JM, Papandonatos GD, Peter I, Huggins GS, Raynor HA, Delahanty LM, Cheskin LJ, Balasubramanyam A, Wagenknecht LE, Wing RR; Genetic Subgroup of Look AHEAD; Look AHEAD Research Group. Obesity susceptibility loci and dietary intake in the Look AHEAD Trial. Am J Clin Nutr. 2012 Jun;95(6):1477-86. doi: 10.3945/ajcn.111.026955. Epub 2012 Apr 18. PMID 22513296